CLINICAL TRIAL: NCT04488848
Title: Effect of Rapid Glucose Excursion Versus Continuous Glucose Infusion on Cardiovascular and Metabolic Parameters in Healthy Volunteers
Brief Title: Cardiometabolic Effects of Rapid Glucose Excursion
Acronym: ERGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barmherzige Brüder Linz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ERGE
Record Dates: First submitted 2019-08-07; First posted 2020-07-28 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Experimental
MeSH Terms: conditions — Diabetes Mellitus, Experimental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continous glucose (Placebo Comparator): continous glucose infusion (60 grams over 3 hours)
  Interventions: Other: continuous clucose
- bolus (excursion) (Experimental): 3 x 20 grams of glucose as a bolus over 6 minutes at t0, 60 minutes and 120 minutes
  Interventions: Other: bolus glucose

INTERVENTIONS:
Other: bolus glucose — bolus Glucose
  Arms: bolus (excursion)
Other: continuous clucose — continuous clucose
  Arms: continous glucose

SUMMARY:
The effects of rapid glucose excursions, induced by intravenous bolus application of glucose in healthy probands, on cardiometabolic and inflammatory parameters will be investigated

DETAILED DESCRIPTION:
BACKGROUND: It is well known that people with diabetes have a five times higher risk of dying of cardiovascular death than non-diabetics. However not only hyperglycaemia per se but also glycaemic variability is currently particularly regarded as a risk factor for cardiovascular and microvascular complications. Intermittent blood sugar excursions with pronounced fluctuations between high and low values instead of constant, even increased blood sugar exposure, have been shown to be more harmful in several studies.

AIM: The aim of this study is to determine the effect of rapid glucose excursion versus continuous glucose infusion on cardiovascular and metabolic parameters in healthy volunteers.

METHODS/DESIGN: In this study, ten healthy male subjects will be studied on two occasions. In a random order the subjects will receive 3 times 20 grams of glucose intravenously as a bolus or, on the other occasion, 60 grams of glucose continuously over 3 hours. Cardiometabolic biomarkers will be analysed serially to analyse the effects of glucose excursions.

PROSPECT: Glycaemic variability may be a crucial factor in the development of diabetic complications, but there is currently a lack of conclusive evidence. The causes and mechanisms of these negative influences on the cardiovascular system due to high glucose variability have not been sufficiently investigated and are therefore not fully understood so far. To date, however, there have been no studies with acutely altered glucose concentrations in healthy volunteers that have investigated the effects on traditional as well as recently identified cardiovascular and metabolic biomarkers. Knowledge of such effects may improve the therapeutic strategy in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years or older with no disease history
* written informed consent

Exclusion Criteria:

* receiving any medication
* probands who suffer from infectious disease

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — homogeneity
Enrollment: 10 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Interleukin-6 | 48 hours
  measurement of the concentration of IL-6 (parameter of inflammation) in the serum over time following infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Barmherzige Brüder Linz - Innere Medizin, Linz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feldbauer R, Heinzl MW, Klammer C, Resl M, Pohlhammer J, Rosenberger K, Almesberger V, Obendorf F, Schinagl L, Wagner T, Egger M, Dieplinger B, Clodi M. Effect of repeated bolus and continuous glucose infusion on a panel of circulating biomarkers in healthy volunteers. PLoS One. 2022 Dec 27;17(12):e0279308. doi: 10.1371/journal.pone.0279308. eCollection 2022. PMID 36574434